CLINICAL TRIAL: NCT00020410
Title: Phase I Study Of Yttrium 90-labeled Monoclonal Antibody B3 With Autologous Stem Cell Support For Metastatic Breast Cancer
Brief Title: Radiolabeled Monoclonal Antibody Followed by Peripheral Stem Cell Transplantation in Treating Patients With Relapsed or Metastatic Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068405; NCI-00-C-0206; NCI-213; NCT00006197 (obsolete NCT alias)
Record Dates: First submitted 2001-07-11; First posted 2003-01-27 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2003-09

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer; male breast cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male | interventions — Filgrastim; Peripheral Blood Stem Cell Transplantation

INTERVENTIONS:
Biological: filgrastim
Procedure: peripheral blood stem cell transplantation
Radiation: yttrium Y 90 monoclonal antibody B3

SUMMARY:
RATIONALE: Radiolabeled monoclonal antibodies can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells. Peripheral stem cell transplantation may allow the doctor to give higher doses of monoclonal antibody therapy and kill more cancer cells.

PURPOSE: Phase I trial to study the effectiveness of radiolabeled monoclonal antibody followed by peripheral stem cell transplantation in treating patients who have relapsed or metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of yttrium Y 90 monoclonal antibody B3 followed by autologous peripheral blood stem cell transplantation in patients with relapsed or metastatic breast cancer.
* Determine the toxicity of this treatment regimen in these patients.
* Determine the clinical response in patients treated with this regimen.

OUTLINE: This is a dose-escalation study of yttrium Y 90 monoclonal antibody B3 (Y90 MOAB B3).

Patients receive filgrastim (G-CSF) subcutaneously (SC) daily beginning 4 days prior to peripheral blood stem cell (PBSC) collection and continuing until the target number of cells is reached.

After PBSC collection, patients receive indium In 111 monoclonal antibody B3 IV over 30-60 minutes once within days -7 to -1 for tumor imaging and then Y90 MOAB B3 IV over 30-60 minutes on day 0. After at least day 7, patients undergo autologous PBSC reinfusion. Patients receive G-CSF SC daily beginning 7 days after PBSC reinfusion and continuing until blood counts recover.

Cohorts of 3-6 patients receive escalating doses of Y90 MOAB B3 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Patients are followed at 1 week, 1 month, and then every 2 months thereafter.

PROJECTED ACCRUAL: A total of 20-30 patients will be accrued for this study within 24-36 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed stage IV breast cancer

  * At least 1 site of relapse or metastatic disease
* Progressive disease after at least 1 prior chemotherapy regimen for metastatic disease

  * One regimen must contain an anthracycline and a taxane as adjuvant therapy or for metastatic disease
  * Prior adjuvant chemotherapy allowed
* Measurable or evaluable disease
* Tumor tissue must express B3 antigen on the surface of more than 30% of tumor cells
* No CNS metastasis
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Sex:

* Male or female

Menopausal status:

* Not specified

Performance status:

* ECOG 0-1

Life expectancy:

* Not specified

Hematopoietic:

* Absolute granulocyte count greater than 2,000/mm^3
* Platelet count greater than 100,000/mm^3

Hepatic:

* Bilirubin normal
* SGOT and SGPT no greater than 2 times upper limit of normal
* PT normal
* Hepatitis B surface antigen negative
* Hepatitis C negative

Renal:

* Creatinine no greater than 1.4 mg/dL

Cardiovascular:

* Ejection fraction at least 45% by MUGA or echocardiogram

Pulmonary:

* FEV_1 greater than 60% of predicted
* FVC at least 55% of predicted
* DLCO at least 55% of predicted

Other:

* No known seizure disorders
* No history of autoimmune disease
* No other active malignancy except previously treated basal cell skin cancer
* No other concurrent medical or psychiatric condition that would preclude study participation
* HIV negative
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Chemotherapy
* No prior mouse antibody

Chemotherapy:

* See Disease Characteristics
* At least 4 weeks since prior chemotherapy (6 weeks for mitomycin or nitrosoureas) and recovered
* No prior high-dose chemotherapy with bone marrow or stem cell transplantation

Endocrine therapy:

* At least 4 weeks since prior hormonal therapy
* No concurrent chronic steroids

Radiotherapy:

* At least 4 weeks since prior local radiotherapy to one site and recovered
* No prior radiotherapy to the pelvis and/or spine

Surgery:

* Not specified

Other:

* No concurrent anticoagulants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-02

CONTACTS AND LOCATIONS:
Overall Officials: Claude Sportes, MD, Study Chair — National Cancer Institute (NCI)
Locations (2):
- United States (2):
  - Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland
  - Center for Cancer Research, Bethesda, Maryland